CLINICAL TRIAL: NCT03770767
Title: A Randomised Controlled Trial Comparing the Effect of the Faster-acting Insulin Analog - Insulin Fiasp® - Versus Insulin Novorapid® in the Treatment of Women With Type 1 or Type 2 Diabetes During Pregnancy and Lactation. The Copen-fast Trial
Brief Title: Insulin Fiasp vs. Insulin Novorapid During Pregnancy and Laction in Women With Pre-existing Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Lene Ringholm, Chief physician, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111
Record Dates: First submitted 2018-12-06; First posted 2018-12-10 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Diabetes Mellitus; Pregnancy Complications
MeSH Terms: conditions — Diabetes Mellitus; Pregnancy Complications

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention with insulin Fiasp (Experimental): Women randomized to insulin Fiasp
  Interventions: Drug: Faster-acting Aspart insulin Fiasp
- Control (insulin Novorapid) (Active Comparator): Women randomized to insulin NovoRapid
  Interventions: Drug: Control (insulin Novorapid)

INTERVENTIONS:
Drug: Faster-acting Aspart insulin Fiasp — Randomization to treatment with insulin Fiasp
  Other Names: Insulin Fiasp
  Arms: Intervention with insulin Fiasp
Drug: Control (insulin Novorapid) — Randomization to standard treatment with insulin Novorapid
  Other Names: First generation insulin analog
  Arms: Control (insulin Novorapid)

SUMMARY:
A randomised controlled, open-label trial in an unselected cohort of pregnant women with type 1 or type 2 diabetes allocated to insulin Fiasp® or insulin NovoRapid® during pregnancy and lactation.

ELIGIBILITY:
Inclusion criteria

* Women, age ≥ 18 years
* Duration of type 1 diabetes (or mature onset of diabetes in the young) ≥ 12 months
* Type 2 diabetes (any duration)
* Pregnant with an intrauterine singleton living fetus confirmed by an ultrasound scan between 8+0 and 13+6 gestational weeks
* Routine use of insulin pump therapy, insulin detemir, insulin degludec, insulin glargine, insulin abasaglar, insulin toujeo or Neutral Protamine Hagedorn insulin and willing to continue routine treatment modality
* Women with type 1 diabetes using an insulin pump compatible with trial products
* Women with type 2 diabetes treated with diet, oral antidiabetic therapy or pre-mixed insulin before pregnancy and willing to change to trial medication according to randomization or to an appropriate long-acting insulin analogue, as indicated
* Proficiency in Danish to understand oral and written information

Exclusion criteria

• Severe mental or psychiatric barriers or concurrent disease on the decision of the principal investigator

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Birth weight standard deviation score | At delivery
  Offspring birth weight (measured as standard deviation score) adjusted for gestational age and gender

SECONDARY OUTCOMES:
HbA1c levels | At inclusion in early pregnancy, at 21 weeks in pregnancy, at 33 weeks in pregnancy, at 36 weeks in pregnancy, at 1 month after delivery, at 3 months after delivery
  HbA1c levels in pregnancy, one and three months after delivery
Postprandial self-monitoring of plasma glucose (SMPG) levels | 9 months
  Postprandial self-monitoring of plasma glucose (SMPG) levels in pregnancy
Preprandial self-monitoring of plasma glucose (SMPG) levels | 9 months
  Preprandial self-monitoring of plasma glucose (SMPG) levels in pregnancy
Insulin treatment and dose (IU) including insulin pump settings | At inclusion in early pregnancy, at 21 weeks in pregnancy, at 33 weeks in pregnancy, at 36 weeks in pregnancy, at 1 month after delivery, at 3 months after delivery
  Type of insulin, dose (IU) during pregnancy, around delivery and until 3 months after delivery. In women on insulin pump therapy: appropriate insulin pump dosing (IU) during pregnancy, around delivery and until 3 months after delivery.
Continuous glucose monitoring data | 9 months
  The amount of time during CGM use spent in the target range 3.5-7.8 mmol/l, with glucose <3.5 mmol/L and glucose >7.8 mmol/L at night-time (23 pm to 7 am) and over 24 h, respectively, in pregnancy and around delivery (in the morning for induction of labour or planned caesarean section). • The percentage of time during the first one-week period after delivery spent in the target range 3.9-10.0 mmol/L, with glucose <3.9 mmol/L and glucose >10.0 mmol/L at night-time (23 pm to 7 am) and over 24 h, respectively.
Severe hypoglycemia | 2 years
  The incidence of severe hypoglycemia in the year preceding pregnancy, during pregnancy and the first three months after giving birth
Mild hypoglycaemia | 12 months
  The incidence of mild hypoglycemia during pregnancy and the first three months after giving birth.
Maternal weight | At inclusion in early pregnancy, at 21 weeks in pregnancy, at 33 weeks in pregnancy, at 36 weeks in pregnancy, at 1 month after delivery, at 3 months after delivery
  Maternal weight in pregnancy and after delivery
Pregnancy complications and outcomes | 9 months
  The prevalence of miscarriage, mode of delivery, early preterm delivery (before 34 completed weeks), preterm delivery (before 37 completed weeks), preeclampsia and perinatal death
Fetal overgrowth | At birth
  The prevalence of fetal overgrowth, defined as the offspring birth weight SD score +1.28 or >90th percentile
Infant weight | 3 months
  Infant weight during the first 3 months of life
Neonatal morbidity (neonatal hypoglycaemia, jaundice, respiratory distress and duration of stay in neonatal intensive care unit) and infant morbidity evaluated as hospitalization during the first 3 months of life (after discharge in the neonatal period) | 3 months
  Neonatal morbidity

CONTACTS AND LOCATIONS:
Overall Officials: Lene Ringholm, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Center for Pregnant Women with Diabetes, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Baseline data can be shared upon request.

REFERENCES:
- [Derived] Norgaard SK, Soholm JC, Mathiesen ER, Norgaard K, Clausen TD, Holmager P, Do NC, Damm P, Ringholm L. Faster-acting insulin aspart versus insulin aspart in the treatment of type 1 or type 2 diabetes during pregnancy and post-delivery (CopenFast): an open-label, single-centre, randomised controlled trial. Lancet Diabetes Endocrinol. 2023 Nov;11(11):811-821. doi: 10.1016/S2213-8587(23)00236-X. Epub 2023 Oct 4. PMID 37804858
- [Derived] Norgaard SK, Mathiesen ER, Norgaard K, Ringholm L. Comparison of Glycemic Metrics Measured Simultaneously by Intermittently Scanned Continuous Glucose Monitoring and Real-Time Continuous Glucose Monitoring in Pregnant Women with Type 1 Diabetes. Diabetes Technol Ther. 2021 Oct;23(10):665-672. doi: 10.1089/dia.2021.0109. Epub 2021 Jun 25. PMID 34086494
- [Derived] Norgaard SK, Mathiesen ER, Norgaard K, Clausen TD, Damm P, Ringholm L. CopenFast trial: Faster-acting insulin Fiasp versus insulin NovoRapid in the treatment of women with type 1 or type 2 diabetes during pregnancy and lactation - a randomised controlled trial. BMJ Open. 2021 Apr 9;11(4):e045650. doi: 10.1136/bmjopen-2020-045650. PMID 33837106